CLINICAL TRIAL: NCT01593293
Title: A Randomized, Open-label, Phase III Study Comparing Pemetrexed With and Without Carboplatin in Elderly Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Pemetrexed With or Without Carboplatin for Elderly Non-squamous Non-small Cell Lung Cancer
Acronym: ACE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Eli Lilly and Company (Industry); Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Sang-We Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC 2011-0857; AMC 2011-0857 (Other: Asan Medical Center)
Record Dates: First submitted 2012-01-11; First posted 2012-05-08 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Elderly patients; Non-squamous Non-small Cell Lung Cancer; Pemetrexed; Carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PemCarbo (Active Comparator): Pemetrexed/Carboplatin arm
  Interventions: Drug: PemCarbo
- Pem only (Active Comparator): Pemetrexed arm
  Interventions: Drug: Pem only

INTERVENTIONS:
Drug: PemCarbo — Pemetrexed 500mg/m2, Carboplatin AUC5 intravenously q 3 weeks for 4 cycles, followed by pemtrexed 500mg/m2 q 3 weeks for maintenance therapy
  Other Names: Alimta: brand name of Pemetrexed
  Arms: PemCarbo
Drug: Pem only — Pemetrexed 500mg/m2 intrvenously q 3 weeks till progression or unacceptable toxicity.
  Other Names: Alimta: brand name of pemetrexed
  Arms: Pem only

SUMMARY:
The number of NSCLC patients above 70 years of age who are non-squamous histology is increasing around the world. Although previous guidelines often recommend single agent therapy for NSCLC, recent studies suggest that platinum doublets may be better than standard monotherapy in elderly. We hypothesize that for elder patients (≥70 years of age) with non-squamous NSCLC, pemetrexed and carboplatin is more effective than pemetrexed monotherapy in terms disease progression, overall survival, and quality of life and tolerability.

DETAILED DESCRIPTION:
The treatment of NSCLC in elderly has been subject to discussion for years. While platinum doublets consisting of cisplatin or carboplatin and another cytotoxic agent demonstrate a survival advantage compared with single agents generally, evidence of treatment efficacy for patients with diminished performance status (PS) or with age older than 70 years is limited. Guidelines from the US and Europe have preferred single-agent chemotherapy for the elderly and PS 2 patients. However, increasing studies are exploring this issue and presenting data that favour doublet therapy. The addition of carboplatin to paclitaxel and cisplatin to docetaxel have shown evidence that patients over 70 benefit more in face of increased toxicities.

This study is designed to be multi-center, open-label, prospective, randomized, two-arm, parallel, phase III trial of elderly patients(≥70 years old) with metastatic non-squamous NSCLC (Stage IV by AJCC 7th) who have not received prior systemic chemotherapy or biological therapy. Approximately 266 patients will be enrolled into the trial. This study compares the doublet therapy of pemetrexed (500 mg/m2) and carboplatin (AUC 5 mg/mL*min) administered intravenously every 21 days for 4 cycles followed by pemetrexed (500 mg/m2) every 21 days for maintenance therapy (Arm A) to single therapy of pemetrexed (500 mg/m2) every 21 days till progression or unacceptable toxicity (Arm B). Pemetrexed will be administered with vitamin B12 and folate supplements.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced non-squamous non-small cell lung cancer (stage IV, AJCC 7th)
* Age 70 years old or older
* Eastern Cooperative Oncology Group performance status 0-1
* Measurable or assessable disease as defined by RECIST 1.1
* Estimated life expectancy of more than 3 months
* Adequate bone marrow function(Absolute Neutrophil Count (ANC) ≥ 1,500/µL, platelets ≥ 100,000/µL, hemoglobulin ≥ 9 g/dL)
* Adequate renal function: creatinine < 1 x upper normal limit (UNL) or creatinine clearance(Ccr) using Cockroft and Gault formula ≥45 ml/min
* Adequate hepatic function: bilirubin < 1.5 x UNL, AST/ALT levels < 3 x UNL, alkaline phosphatase < 3 x UNL (except in case of bone metastasis without any liver disease)
* Written informed consent

Exclusion Criteria:

* Prior systemic chemotherapy or biological therapy
* Contraindication to any drug contained in the chemotherapy regimen
* Clinically significant third-space fluid collections (e.g. pleural effusion and pericardial effusion) that cannot be controlled by drainage or other procedures prior to study enrollment
* Active infection which would compromise the patient's ability to tolerate treatment
* Requirement for major surgery within 4 weeks of study entry
* Myocardial infarction, uncontrolled arrhythmias, symptomatic angina pectoris, cardiac failure within the previous 6 months
* Unable to discontinue administration of aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs); Aspirin or NSAIDs should be at least 5 days before pemetrexed administration
* Presence or history of CNS metastasis (except if adequately treated and is not receiving steroid therapy for at least 2 weeks; at least 2 weeks for whole brain radiation or at least 1 week for gamma knife surgery)
* Peripheral neuropathy ≥ grade 2
* History of another malignancy within the last five years except cured basal cell carcinoma of skin, cured carcinoma in-situ of uterine cervix and cured thyroid malignancy
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Other serious illness or medical conditions

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | The study lasts for 30 months of which subject accrual occurs in the first 24 months
  To compare the progression free survival of elderly patients (≥70 years old) with non-squamous NSCLC receiving doublet of carboplatin and pemetrexed to patients receiving pemetrexed alone.

SECONDARY OUTCOMES:
Objective response rate, Overall survival, Safety and Quality of life | The study lasts for 30 months of which subject accrual occurs in the first 24 months
  1. To compare the following efficacy variables between treatment arms:
     * Objective response rate
     * Overall survival
  2. To compare the safety and adverse event profile between treatment arms
  3. To assess the impact of treatment on patient-rated quality of life (FACT-L)

CONTACTS AND LOCATIONS:
Overall Officials: Sang-We Kim, M.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea